CLINICAL TRIAL: NCT01439841
Title: The Effect of Probiotics on Microbial Translocation and Immune Activation in HIV-1 Infection. A Randomised Placebo-controlled Trial
Brief Title: The Effect of Probiotics in HIV-1 Infection
Acronym: ProGut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Karolinska University Hospital (Other); Tine (Industry)
Responsible Party: Principal Investigator, MariusTrøseid, Marius Trøseid, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ProGut1.0
Record Dates: First submitted 2011-09-16; First posted 2011-09-23 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: HIV-1 Infection
Keywords: HIV; microbial translocation; immune activation; probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotics (Experimental): A multi-strain Probiotic consisting of Lactobacillus rhamnosus GG, Lactobacillus acidophilus La-5 and Bifidobacterium animalis subsp. lactis Bb-12 added to fermented skimmed milk (Biola®, TINE SA, Oslo), 250 mL/day for 8 weeks.
  Interventions: Dietary Supplement: Multi-strain probiotic
- Placebo (Placebo Comparator): Fermented and subsequently heat-treated, sterile skimmed milk (TINE SA) as active placebo.
  Interventions: Dietary Supplement: Placebo
- Control (No Intervention): No intervention

INTERVENTIONS:
Dietary Supplement: Multi-strain probiotic — The product consists of Lactobacillus rhamnosus GG, Lactobacillus acidophilus La-5 and Bifidobacterium animalis subsp. lactis Bb-12 added to fermented skimmed milk
  Other Names: Brand name Biola®
  Arms: Probiotics
Dietary Supplement: Placebo — Fermented and subsequently heat-treated, sterile skimmed milk
  Arms: Placebo

SUMMARY:
HIV progression is closely associated with chronic immune activation driven by leakage of bacterial products from a damaged gut, the investigators largest immunological organ. Notably, the degree of immune activation has been suggested to be a better predictor of disease progression than plasma viral load, and markers of immune activation and gut damage have been identified as therapeutic targets per se. The major damage by HIV to the immune system is an initial massacre of gut mucosal CD4+ Th17 cells. Interestingly, a normal gut flora has been shown to induce the maturation of Th17 cells in the small intestine mucosa. Preliminary reports have shown that the gut flora is altered in HIV-1 infection compared to controls. In this project, the investigators will characterize microbial composition of gut flora in chronic HIV infection with ultradeep sequencing. Gut flora composition will be related to clinical data as well as quantitative data of circulating microbial products and activation markers. Second, in a randomized clinical trial (RCT) the effect of probiotic lactobacilli on HIV pathogenesis and progression will be tested. This Gram-positive strain is clinically tested and is able to colonize the gut.

DETAILED DESCRIPTION:
Objectives:

To explore (i) the safety and tolerability, and (ii) the efficacy of probiotics on HIV-associated microbial translocation, systemic immune activation, disease progression and composition of gut microbiota in chronic HIV-1 infection.

Methodology/Study design:

Approximately 50 patients without current indication for antiretroviral treatment (ART) and 50 patients receiving ART without normalised CD4 counts will be included. A controlled clinical trial will be carried out within each stratum randomised in a 2:1:1 fashion to double blinded intervention and placebo arms as well as an open, untreated control arm, respectively.

ELIGIBILITY:
Inclusion Criteria:

* For patients without ART: Confirmed diagnosis of HIV infection > 6 months and CD4+ T cell count < 900
* For patients on stable, effective ART: HIV RNA < 50 copies/ml > 6 months and CD4+ T cell count > 500
* Signed informed consent.

Exclusion Criteria:

* Severe illness requiring hospitalization
* Systemic antibiotics or probiotics the last two months
* Current immune modulating therapy
* Infectious diarrhea
* Inflammatory bowel disease
* Acute primary HIV infection
* Patients immigrating from Africa, Asia or Latin-America within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety | 2 months
  Adverse events monitoring during the study period of 2 months
Changes in measures of microbial translocation | 2 months
  Changes in plasma leves of lipopolysaccharide (LPS) and soluble CD14 from baseline to 2 months (end of study)
Changes in markers of immune activation | 2 months
  Changes in CD38, HLA-DR and PD-1 on CD8+ and CD4+ T cells from baseline to 2 months (end of study)

SECONDARY OUTCOMES:
Disease progression in untreated patients | 2 months
  Changes in CD4 count, viral load, clinical events and indication for ART from baseline to 2 months (end of study)
Immune reconstitution in ART treated patients | 2 months
  Changes in CD4 count from baseline to 2 months (end of study)
Gut microbiota composition | 2 months
  Changes in gut microbiota (454 pyrosequencing of fecal samples) from baseline to 2 months (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Gokstad, MD, PhD, Study Director — Oslo University Hospital; Marius Trøseid, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Oslo University Hospital, Oslo, Norway
- Karolinska University Hospital Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Stiksrud B, Nowak P, Nwosu FC, Kvale D, Thalme A, Sonnerborg A, Ueland PM, Holm K, Birkeland SE, Dahm AE, Sandset PM, Rudi K, Hov JR, Dyrhol-Riise AM, Troseid M. Reduced Levels of D-dimer and Changes in Gut Microbiota Composition After Probiotic Intervention in HIV-Infected Individuals on Stable ART. J Acquir Immune Defic Syndr. 2015 Dec 1;70(4):329-37. doi: 10.1097/QAI.0000000000000784. PMID 26258571